CLINICAL TRIAL: NCT04285814
Title: Technology Development for Noninvasive Prenatal Genetic Diagnosis Using Whole Fetal Cells From Maternal Peripheral Blood
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Baylor College of Medicine (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ronald J Wapner, MD, Vice Chair, Research, OBGYN, Columbia University
Other Study IDs: AAAS9107; 3R01HD055651 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Copy Number Abnormality; Prenatal Diagnosis; Genetic Disease
Keywords: noninvasive prenatal testing; microarray; fetal cells; prenatal diagnosis
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Remaining blood samples and products (including DNA) will be stored for future research on WFC testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal CMA: 150 women whose blood samples will be drawn for WFC testing who previously had a CMA performed with normal results.
  Interventions: Diagnostic Test: Whole Fetal Cell (WFC) Testing
- Abnormal CMA: 150 women whose blood samples will be drawn for WFC testing who previously had a CMA performed with abnormal results.
  Interventions: Diagnostic Test: Whole Fetal Cell (WFC) Testing

INTERVENTIONS:
Diagnostic Test: Whole Fetal Cell (WFC) Testing — Performing WFC testing on blood specimens.

SUMMARY:
Amniocentesis (amnio) and chorionic villus sampling (CVS) can reliably detect many smaller DNA/genetic abnormalities that cannot be reliably diagnosed by cell-free noninvasive prenatal testing (NIPT) that is in widespread use. The investigators present evidence that a cell-based form of NIPT, here called Single Fetal Cell (SFC) testing, using a blood sample from the mother can detect most or all of the genetic abnormalities that are detected using amnio or CVS. This study proposes to compare the effectiveness of SFC testing in detecting abnormalities already detected by amnio or CVS in women already undergoing these tests as part of their clinical care because of fetal ultrasound abnormalities.

DETAILED DESCRIPTION:
This is a revision to a project entitled "Prenatal Genetic Diagnosis by Genomic Sequencing: A Prospective Evaluation." This study proposes to test the utility and accuracy of a new form of cell-based noninvasive prenatal testing (NIPT), here called noninvasive Single Fetal Cell (SFC) testing. After many years of development work, the researchers published evidence for the feasibility of SFC testing in 2016. Extensive recent preliminary data show considerable improvements in SFC testing. Current forms of cell-free NIPT testing do not provide reliable detection of medium to smaller size deletions and duplications that cause a variety of genetic disabilities. Preliminary data indicate that SFC testing using fetal trophoblasts from mother's blood can detect aneuploidy and subchromosomal deletions and emphasize the importance of analyzing single cells, since some fetal cells are apoptotic and some are in S phase of the cell cycle replicating their DNA. Both apoptosis and S phase interfere with copy number analysis in differing ways, and pooling cells prior to barcoding individual cells results in loss of data quality. Preliminary data from two pilot validation studies demonstrate that reliable data can be collected on the large majority of patients, although data on this point would be greatly expanded by this project.

Preliminary data show very robust detection of all aneuploidies and clear definition of genomic deletions as small as 1 Mb and duplications as small as 1.5 Mb. The first aim is to perform blinded SFC testing on 50 cases per year with congenital anomalies with abnormal karyotype or chromosomal microarray (CMA) and 50 cases per year with congenital anomalies and normal CMA. This will provide a direct measure of success rate and the false positive and false negative rates for SFC testing compared to CMA. The second aim will be to use the WGA products and frozen unamplified cells available from aim 1 to further improve SFC testing to include targeted detection of inherited or de novo pathogenic point mutations in the cases undergoing WGS as part of the parent grant, confirmation of very small CNVs detected by WGS, restudy of false positive or false negative results from aim 1, and in the future could attempt to perform genome wide detection of de novo mutations. Capitalizing on the resources available through the parent grant, there is the opportunity to test whether SFC testing has the potential to transform genetic prenatal diagnosis so that all genetic changes, whether CNV or point mutation, and whether inherited or de novo, could be detected even in low risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Have already had a CVS or amniocentesis (blood sample collected >= 7 days after procedure).
* Have already received an abnormal (case) or normal (control) CMA/karyotype/FISH result from the CVS or amniocentesis.

Exclusion Criteria:

* Unavailability of maternal blood sample at least 7 days post-procedure.
* Language barrier (non-English or Spanish speaking and no adequate interpreter)
* Maternal age of less than 18 years
* Higher order multiple pregnancy (triplet or greater)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be pregnant women.
Study Population: Pregnant women presenting at the study sites who have a karyotype and/or CMA performed will be recruited for this study. Half of the women will have a normal CMA (150) and half will have an abnormal CMA (150).
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Using a population of pregnancies with abnormal and normal karyotypes and CMAs, determine the false positive, false negative, true positive, and true negative rates of WFC testing. | 3 years
Determine the technical success rate for WFC testing including number of scorable cells for each sample. | 3 years
Determine the level of resolution for detecting deletions/duplications by WFC testing based on "spiked in" samples of known CNVs and on analysis of naturally occurring CNVs in fetal cells. | 3 years
Determine capability and success rate for genotyping single gene mutations including de novo and inherited single gene mutations and benign SNPs. | 3 years

SECONDARY OUTCOMES:
Evaluate WFC testing results according to gestational age at testing, specific anomalies, maternal weight, and multiple gestations. | 3 years
Determine whether cells are more frequent in pregnancies resulting in adverse pregnancy outcomes including preeclampsia. | 3 years
Improve methods for genotyping single cells including ability to perform genotyping and genome-wide copy number analysis on the same cell. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wapner, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
The project dataset and associated genomic data be widely shared with the scientific community for research through the controlled access dbGAP repository or comparable databases while carefully observing standards of patient privacy, confidentiality, and management of health information complying with the NIH Genomic Data Sharing policy. The data-sharing of genetic data will be in dbGaP. Data will be generated in all years of the study and submitted at study completion. Resources including study protocols, informed consent templates, result report templates and bioinformatic tools will also be made available through open access databases and public web sites. We will make datasets and informatics tools available through approved platforms for sharing with the larger scientific community. We will store remaining DNA samples with permission to use these samples for future research related to WFC. These specimens will be stored in a coded fashion.